CLINICAL TRIAL: NCT01657526
Title: An Observer-blind Study to Evaluate the Safety, Reactogenicity and Immunogenicity of GSK Biologicals' Non-typeable Haemophilus Influenzae (NTHi) Investigational Vaccine (GSK2838497A) in Healthy Adults
Brief Title: Safety, Reactogenicity and Immunogenicity of GlaxoSmithKline (GSK) Biologicals' Non-typeable Haemophilus Influenzae (NTHI) Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 116018
Record Dates: First submitted 2012-08-02; First posted 2012-08-06 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Respiratory Disorders
Keywords: Healthy adults; Safety; Reactogenicity; Immunogenicity; Non-typeable H. Influenzae (NTHi)
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- Group A (Experimental): Subjects in this group will receive GSK Biologicals' NTHi candidate vaccine in Step 1 of the study
  Interventions: Biological: GSK Biologicals' Non-Typeable H. influenzae (GSK2838500A)
- Group B (Placebo Comparator): Subjects in this group will receive placebo in Step 1 of the study
  Interventions: Biological: Saline placebo
- Group C (Experimental): Subjects in this group will receive GSK Biologicals' NTHi candidate vaccine in Step 2 of the study
  Interventions: Biological: GSK Biologicals' Non-Typeable H. influenzae (GSK2838501A)
- Group D (Placebo Comparator): Subjects in this group will receive placebo in Step 2 of the study
  Interventions: Biological: Saline placebo

INTERVENTIONS:
Biological: GSK Biologicals' Non-Typeable H. influenzae (GSK2838500A) — Administered intramuscularly (IM) in the deltoid region of non-dominant arm
  Arms: Group A
Biological: GSK Biologicals' Non-Typeable H. influenzae (GSK2838501A) — 2 doses administered IM in the deltoid region of non-dominant arm
  Arms: Group C
Biological: Saline placebo — 2 doses administered IM in the deltoid region of non-dominant arm
  Arms: Group B; Group D

SUMMARY:
The purpose of this study is to evaluate the safety, reactogenicity and immunogenicity of GSK Biologicals' NTHi candidate vaccine in adults, administered for the first time in humans.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject.
* A male or female between, and including, 18 and 40 years of age at the time of the first vaccination.
* Healthy subjects as established by medical history, physical examination and laboratory assessment before entering into the study.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccines within 30 days preceding the first dose of study vaccines, or planned use during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product.
* Planned administration/administration of a vaccine/product not foreseen by the study protocol in the period starting 30 days before the first vaccine dose and ending 30 days after the last dose of vaccines.
* Previous vaccination with a vaccine containing NTHi antigens.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose, or equivalent. Topical steroids are allowed.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the first dose of study vaccines or planned administration during the study period.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Laboratory evidence of clinically significant haematological (complete blood cell count [Red Blood Cells (RBC), White Blood Cells (WBC)], WBC differential count, platelets count and haemoglobin level) and biochemical (Alanine Aminotransferase [ALT], Aspartate Aminotransferase [AST], creatinine and lactate dehydrogenase [LDH]) abnormalities as per the opinion of the investigator based on the local laboratory normative data.
* Acute disease and/or fever at the time of enrolment.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* History of or current condition preventing intramuscular injection as bleeding or coagulation disorder.
* Malignancies within previous 5 years (excluding non-melanic skin cancer) and lymphoproliferative disorders.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* History of chronic alcohol consumption and/or drug abuse.
* Any other condition that the investigator judges may interfere with study findings.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2012-08-08 (Actual); Primary Completion 2013-11-25 (Actual); Study Completion 2013-11-25 (Actual)

PRIMARY OUTCOMES:
Occurrence of solicited local and general adverse event (AE), in all subjects, in all vaccine groups | During a 7-day follow-up period (i.e. day of vaccination and 6 subsequent days) after each vaccination.
Occurrence of any unsolicited AE, in all subjects, in all vaccine groups | During a 30-day follow-up period (i.e. day of vaccination and 29 subsequent days) after each vaccination.
Occurrence of haematological and biochemical laboratory abnormalities, in all subjects, in all vaccine groups | At baseline (Screening visit) and after each vaccination.
Occurrence of any serious adverse event (SAE), in all subjects, in all vaccine groups | From first vaccination to study conclusion (Day 420).
Occurrence of any potential Immune-Mediated Disease (pIMDs) in all subjects, in all vaccine groups | From first vaccination to study conclusion (Day 420).

SECONDARY OUTCOMES:
Humoral immune response to components of the NTHi vaccine formulations, in all subjects, in all vaccine groups | Prior to each vaccination and 30 days post each vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Adelaide, South Australia, Australia

REFERENCES:
- See also: Results for study 116018 can be found on the GSK Clinical Study Register — https://www.gsk-clinicalstudyregister.com/study/116018?search=study&b%22b''%22#rs